CLINICAL TRIAL: NCT03404895
Title: The Mount Sinai Diabetic Foot Ulcer Prospective Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Windsor Ting (Other)
Responsible Party: Sponsor-Investigator, Windsor Ting, Associate Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GCO 17-2608
Record Dates: First submitted 2018-01-12; First posted 2018-01-19 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Diabetes; Diabetic Foot Ulcer; Edema
Keywords: DFU; Vein; Stent
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Foot; Edema

STUDY DESIGN:
Intervention Model Description: Subjects are randomized in the OR to one of two study arms: conventional therapy vs. conventional therapy + venous stent(s).
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Conventional Therapy (Sham Comparator): Conventional therapy of DFU comprises of four components: local wound care, antibiotic therapy, debridement and amputation, and pressure offloading.
  Interventions: Device: Conventional Therapy
- Conventional Therapy + venous stent(s) (Active Comparator): Patients will receive a venous stent in addition to conventional therapy
  Interventions: Device: Conventional Therapy; Device: Venous Stent(s)

INTERVENTIONS:
Device: Conventional Therapy — Local wound care consists of at least once daily dressing Occasionally, a limited bedside debridement is indicated to excise small quantity of devitalized tissues and to provide better drainage. Antibiotic therapy including both gram-positive and gram-negative coverage when the DFU appears infected is guided by wound cultures and when necessary, Infectious Disease consultation. Debridement and amputation will be performed as clinically indicated. To promote healing after the more acute processes have been addressed, pressure offloading is frequently helpful in the healing of DFU. Pressure offloading treatment ranges from special dressings and devices to special diabetic foot wares. Offloading will be utilized as indicated.
Device: Venous Stent(s) — After PVOO is confirmed by venography and IVUS, and patient subject is randomized to conventional therapy and stent placement, stent placement is performed immediately at the same sitting.
  Arms: Conventional Therapy + venous stent(s)

SUMMARY:
The purpose of this study is to evaluate whether placing stent(s) for a blockage in a leg vein will help improve the healing of diabetic foot ulcers (DFU). The investigators know from having taken care of many patients with diabetic foot ulcers that it is a major cause of disability and amputation. These diabetic foot ulcers frequently heal slowly or not at all. They sometimes become infected and require antibiotic therapy, debridement and amputation. The investigators normally take care of a diabetic foot ulcer with a combination of local wound care, surgical debridement if necessary, antibiotics if there is an infection, and reduction of pressure on the area of the foot with the ulcer. The investigators observed that some patients with a diabetic foot ulcer also have a blockage in a major leg vein referred to as the iliac vein. This blockage in the iliac vein prevents the proper flow of blood from the leg. This blockage results in pressure within the leg veins leading to swelling in the legs which may also prevent healing of the diabetic foot ulcer. This study will investigate whether placing stent(s) to treat the blockage(s) will improve healing of the diabetic foot ulcer and reduce some of the complications associated with a diabetic foot ulcer. The results of this study could result in a new treatment that will allow future patients with diabetic foot ulcers to heal better. Right now, placing stents for these blockages in the iliac vein is not the standard of care treatment for a diabetic foot ulcer. In order for us to determine whether stent placement is helpful, the researchers will have to randomize each patient. In other words, to reduce bias, patients will be assigned either to a group receiving a stent or to a group not receiving a stent. Every patient in both groups will receive the standard of care for a diabetic foot ulcer and undergo an x-ray with contrast and intravenous ultrasound examination of the legs. The standard of care for a diabetic foot ulcer may include local wound care, antibiotic therapy, debridement and/or amputation, and pressure offloading in the foot.

DETAILED DESCRIPTION:
This will be a single center, patient-blinded, randomized controlled trial. In the event that a patient does not meet inclusion criteria after signing the consent for and undergoing venogram/IVUS (screen fail), additional patients will be enrolled until 60 patients have been successfully randomized. Up to 80 patients will be consented in order to account for potential screen fails. Randomized patients will be followed monthly until their ulcer heals, every 3 months after healing for one year postoperatively.

Every patient subject will undergo venogram & IVUS. The investigator experience with over 600 patients who underwent venous stenting at Mount Sinai - all of whom had preoperative MR venogram or CT venogram - revealed that pre-operative imaging missed the diagnosis of PVOO in approximately 10% of patients (this is unpublished data). Due to the small sample size of this pilot study, the very low risks associated with venogram and IVUS, and the 100% accuracy of venogram and IVUS in diagnosing PVOO, every study subject will undergo these two imaging studies. Once the diagnosis of PVOO is confirmed, the study subject will be immediately randomized in the OR. Study subjects randomized to convention therapy plus venous stents will undergo venous stent placement at the same sitting. For study subjects randomized to conventional therapy alone, the procedure will be terminated after venogram and IVUS.

ELIGIBILITY:
Inclusion Criteria:

* Presence of diabetic foot ulcer within the foot (located distal to the ankle and proximal to base of toes)
* Lower extremity edema
* MRA or CTA showing stenosis of iliac vein or indirect findings that suggest presence of iliac vein stenosis (distal venous dilation and presence of collateral veins)
* At least one palpable pedal pulse or ABI>0.9 IVUS confirmation of iliac vein stenosis

Exclusion Criteria:

* Previous vein stent implantation involving study leg or inferior vena cava
* Previous bypass surgery or endovascular intervention involving study leg
* Known metal allergy
* Known reaction or sensitivity to iodinated contrast that cannot be managed with premedication
* Acute deep venous thrombosis involving either leg
* Known history of chronic occlusion of any vein in the study leg
* Venous compression caused by tumor encasement
* Venous outflow obstruction caused by tumor thrombus
* Elevated baseline blood creatinine (>1.5)
* Pregnancy
* Life expectancy <12 months

Ages: 30 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-04-13 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Number of days to ulcer healing | average of 1 year
  All patient subjects with an active ulcer will be followed until healing of the ulcer.

SECONDARY OUTCOMES:
Number of subjects whose DFU persisted | 12 months
  Number of subjects whose DFU persisted 12 months post-randomization
Number of recurrent DFU | 12 months
  Number of subjects who had recurrent DFU 12 months post-randomization
Total number of subjects with limb loss | 12 months
  Number of subjects who had limb loss within 12 months post-randomization
Total number of subjects with minor and major amputations | 12 months
  Number of subjects who had major or minor amputations within 12 months post-randomization

CONTACTS AND LOCATIONS:
Overall Officials: Windsor Ting, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided